CLINICAL TRIAL: NCT01111357
Title: Study of HLA Polymorphisms in French West-Indian Patients With Rheumatoid Arthritis : A Case Control Study
Brief Title: Study of Human Leukocyte Antigen (HLA) Polymorphisms in Patients With Rheumatoid Arthritis
Acronym: HLAPRPA
Status: Completed | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: JEAN - BAPTISTE Georges, Service de Rhumathologie CHU de Fort-de-France
Other Study IDs: 09/B/02
Record Dates: First submitted 2010-01-29; First posted 2010-04-27 (Estimated); Last update posted 2010-12-21 (Estimated); Status verified 2010-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Rheumatoid Arthritis according to ACR criteria of diagnosis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood : collect of 10 ml of peripheric blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Collect of 10 ml of peripheric blood for DNA extraction — After signed written consent, all patients have a clinic exam in order to assess the presence of eligibility criteria (Patient with Rheumatoid Arthritis that fulfil the ACR criteria of diagnosis)
  Other Names: Rheumatoid Arthritis; French West-Indian Patients with Rheumatoid Arthritis

SUMMARY:
Rheumatoid arthritis (RA), affects between 0.3% and 1.0% of the population, it can lead to progressive joint destruction and severe disability. To date, two RA genetic susceptibility factors have been identified: HLA-DRB1-SE (Shared epitope) and PTPN22 620W alleles. The predictive value of the alleles for diagnosis of RA was previously investigated in cohorts of caucasians patients with early unclassified arthritis that showed restrained association between RA and HLA-SE. Despite the contribution of HLA to the overall genetic risk has been estimated to range from 30% to 50%, it has never been studied in the French west-Indian population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Rheumatoid Arthritis according to ACR criteria
* Come from French West Indies (At least 3 grandparents are African-Caribbean)
* Sign written informed consent

Exclusion Criteria:

* Minor
* Patient with no Rheumatoid Arthritis according to ACR criteria
* Patient does not agree for a genetic study

For the control

Inclusion Criteria:

* Blood donor
* Sign written informed consent
* Patient with no Rheumatoid Arthritis according to ACR criteria
* Come from French West Indies (At least 3 grandparents are African-Caribbean)

Exclusion Criteria:

* Minor
* Patient does not agree for a genetic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Residents of Martinique with at least 3 African-Caribbean grandparents
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Difference of distribution of HLA alleles in patients and in healthy controls | 1 day

SECONDARY OUTCOMES:
The association between the different HLA alleles among French West-Indian RA patients and the autoantibodies production. | 1 day
The association between the different HLA alleles among French West-Indian RA patients and the radiological damage. | 1 day
The association between the different HLA alleles among French West-Indian RA patients and the response to therapy | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Georges JEAN-BAPTISTE, Professor of medecine, Principal Investigator — CHU de Fort-de-France
Locations (1):
- Service de rhumatologie CHU de Fort-de-France, Fort-de-France, Martinique